CLINICAL TRIAL: NCT02315950
Title: CineMRI/UDS for Evaluating the Physiologic Effect of Botox in Women With Overactive Bladder
Brief Title: The Use of cineMRI to Evaluate Botox in Patients With Medication Refractory Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer T. Anger, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00037210
Record Dates: First submitted 2014-10-28; First posted 2014-12-12 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Other): Botulinum toxin and cineMRI-UDS
  Interventions: Other: Botulinum toxin and cineMRI-UDS

INTERVENTIONS:
Other: Botulinum toxin and cineMRI-UDS — The investigators will be testing the capability of cineMRI combined with simultaneous urodynamics in the context of OAB in this proposal and expect to reveal a new understanding of diseased lower urinary tract physiology. Participants will receive an injection of intravesical botulinum toxin after filling out validated questionnaires and receiving a pre-treatment cineMRI-UDS.

SUMMARY:
With the goal of providing improved treatment to patients with overactive bladder symptoms (OAB), the investigators seek to apply the new technology of time-resolved (cine) MRI combined with urodynamics (UDS) to understand the exact effect of intravesical botulinum toxin on bladder physiology. The investigators will specifically aim to assess the physiological mechanism by which intravesical botulinum alleviates urgency and urge incontinence symptoms in women with OAB refractory to medical therapy.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is defined by the International Continence Society as urinary frequency and urgency, with or without urge urinary incontinence. The burden of OAB on the American public is immense in both human and financial terms. Despite this burden, there is a lack of effective diagnostic and treatment modalities for OAB. Other than two-dimensional video urodynamics, which has remained relatively unchanged for decades, there is a lack of diagnostic modalities that will allow investigators to characterize subtypes of OAB and measure the effects of treatment on bladder physiology. Newer imaging techniques are desperately needed to help guide treatment and predict and improve outcomes of different treatment modalities. Intravesical botulinum toxin is a minimally invasive treatment for OAB refractory to medical therapy. Despite the widespread use of intravesical botulinum toxin injection for OAB refractory to medical therapy, to date the optimal placement of the drug has not been determined. Typically ten injections are given, either dispersed evenly across the bladder or in two rows of five injections. However, it remains unknown which injection method will optimize outcomes and reduce the risk of urinary retention after Botox®. This lack of knowledge is a direct result of the fact that there has been no mechanism to study the effect of Botox® on bladder filling and emptying in a three-dimensional fashion. CineMRI-UDS will provide this mechanism, and has the potential to significantly improve care and urologic education by enhancing the understanding of bladder physiology.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21 years or older
* Overactive bladder symptoms

Exclusion Criteria:

* Age less than 21 years
* Inability to give informed consent
* Claustrophobic

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time-resolved views by CineMRI with urodynamics on overactive bladder physiology | About 10 Months
  CineMRI and urodynamics technology will be used to obtain time-resolved views of the human bladder during filling and voiding. The investigators aim to reveal a new understanding of diseased lower urinary tract physiology during pre and post treatment.

OTHER OUTCOMES:
Improvement in overactive bladder symptoms by smooth muscle paralysis via botulinum toxin injection (100U) | About 10 Months
  This injection is performed under local anesthesia in the office. 100U of botulinum toxin (Botox ®) will be mixed under sterile conditions with 10cc of sterile saline and injected into 10 discrete locations in the bladder. Participants will be asked to fill out questionnaires for the management of clinical and statistical measures.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Anger, MD, MPH, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Beverly Hills, California, United States

REFERENCES:
- [Background] Wein AJ, Rovner ES. Definition and epidemiology of overactive bladder. Urology. 2002 Nov;60(5 Suppl 1):7-12; discussion 12. doi: 10.1016/s0090-4295(02)01784-3. PMID 12493342
- [Background] Lin K, Bi X, Taimen K, Zuehlsdorff S, Lu B, Carr J, Li D. Coronary wall MR imaging in patients with rapid heart rates: a feasibility study of black-blood steady-state free precession (SSFP). Int J Cardiovasc Imaging. 2012 Mar;28(3):567-75. doi: 10.1007/s10554-011-9852-z. Epub 2011 Apr 2. PMID 21461663
- [Background] Zhou X, Rundell V, Liu Y, Tang R, Shah S, Zuehlsdorff S, Li D, Dharmakumar R. On the mechanisms enabling myocardial edema contrast in bSSFP-based imaging approaches. Magn Reson Med. 2011 Jul;66(1):187-91. doi: 10.1002/mrm.22794. Epub 2011 Mar 9. PMID 21394764
- [Background] Tsaftaris SA, Tang R, Zhou X, Li D, Dharmakumar R. Ischemic extent as a biomarker for characterizing severity of coronary artery stenosis with blood oxygen-sensitive MRI. J Magn Reson Imaging. 2012 Jun;35(6):1338-48. doi: 10.1002/jmri.23577. Epub 2012 Jan 13. PMID 22246681
- [Background] Borghesi G, Simonetti R, Goldman SM, Szejnfeld J, Srougi M, Ortiz V, Bruschini H. Magnetic resonance imaging urodynamics. Technique development and preliminary results. Int Braz J Urol. 2006 May-Jun;32(3):336-41; discussion 341. doi: 10.1590/s1677-55382006000300015. PMID 16813681
- [Background] Brubaker L, Richter HE, Visco A, Mahajan S, Nygaard I, Braun TM, Barber MD, Menefee S, Schaffer J, Weber AM, Wei J; Pelvic Floor Disorders Network. Refractory idiopathic urge urinary incontinence and botulinum A injection. J Urol. 2008 Jul;180(1):217-22. doi: 10.1016/j.juro.2008.03.028. Epub 2008 May 21. PMID 18499184
- [Background] Nitti VW, Dmochowski R, Herschorn S, Sand P, Thompson C, Nardo C, Yan X, Haag-Molkenteller C; EMBARK Study Group. OnabotulinumtoxinA for the treatment of patients with overactive bladder and urinary incontinence: results of a phase 3, randomized, placebo controlled trial. J Urol. 2013 Jun;189(6):2186-93. doi: 10.1016/j.juro.2012.12.022. Epub 2012 Dec 14. PMID 23246476
- [Background] Anger JT, Weinberg A, Suttorp MJ, Litwin MS, Shekelle PG. Outcomes of intravesical botulinum toxin for idiopathic overactive bladder symptoms: a systematic review of the literature. J Urol. 2010 Jun;183(6):2258-64. doi: 10.1016/j.juro.2010.02.009. Epub 2010 Apr 18. PMID 20400142
- [Background] Dmochowski R, Chapple C, Nitti VW, Chancellor M, Everaert K, Thompson C, Daniell G, Zhou J, Haag-Molkenteller C. Efficacy and safety of onabotulinumtoxinA for idiopathic overactive bladder: a double-blind, placebo controlled, randomized, dose ranging trial. J Urol. 2010 Dec;184(6):2416-22. doi: 10.1016/j.juro.2010.08.021. Epub 2010 Oct 16. PMID 20952013
- [Background] Jackson S, Donovan J, Brookes S, Eckford S, Swithinbank L, Abrams P. The Bristol Female Lower Urinary Tract Symptoms questionnaire: development and psychometric testing. Br J Urol. 1996 Jun;77(6):805-12. doi: 10.1046/j.1464-410x.1996.00186.x. PMID 8705212
- [Background] Donovan JL, Abrams P, Peters TJ, Kay HE, Reynard J, Chapple C, De La Rosette JJ, Kondo A. The ICS-'BPH' Study: the psychometric validity and reliability of the ICSmale questionnaire. Br J Urol. 1996 Apr;77(4):554-62. doi: 10.1046/j.1464-410x.1996.93013.x. PMID 8777617
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- [Background] Chung SD, Liao CH, Chen YC, Kuo HC. Urgency severity scale could predict urodynamic detrusor overactivity in patients with overactive bladder syndrome. Neurourol Urodyn. 2011 Sep;30(7):1300-4. doi: 10.1002/nau.21057. Epub 2011 May 10. PMID 21560153